CLINICAL TRIAL: NCT04873453
Title: Tolerability and Efficacy of Hemp-Derived CBD for the Treatment of Alcohol Use Disorder
Brief Title: CBD for the Treatment of Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-2694
Record Dates: First submitted 2021-04-20; First posted 2021-05-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Cannabidiol; CBD; Cannabis
MeSH Terms: conditions — Alcoholism; Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full-spectrum Cannabidiol (Active Comparator): 150mg/day of full-spectrum cannabidiol, containing less than 0.3%THC.
  Interventions: Drug: Cannabidiol
- Broad-spectrum Cannabidiol (Experimental): 150mg/day of broad-spectrum cannabidiol, containing 0%THC.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): 150mg/day of hemp-seed oil with no cannabinoids present.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — The current study will directly test the hypothesis that a moderate dose of CBD leads to a reduction in alcohol consumption, alcohol craving, peripheral markers of inflammation, and anxiety.
  Other Names: CBD
  Arms: Broad-spectrum Cannabidiol; Full-spectrum Cannabidiol
Drug: Placebo — Placebo arm
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, parallel group study designed to assess the efficacy of full spectrum cannabidiol (CBD) and broad spectrum CBD, compared to a placebo control (PC), to reduce drinking in participants with moderate alcohol use disorder according to the DSM-V. If eligible for the study, subjects will be randomized to receive one of the conditions for 8 weeks.

DETAILED DESCRIPTION:
The current study will directly test the hypothesis that a moderate dose of cannabidiol (CBD) leads to a reduction in alcohol consumption, alcohol craving, peripheral markers of inflammation, and anxiety. It is further hypothesized that CBD will lead to increased sleep duration and quality among individuals with AUD who want to quit or reduce their drinking. The study will also determine whether the small amount of THC found in full spectrum hemp-derived CBD products produces any negative effects. The hypotheses are grounded in previous studies suggesting that CBD reduces the reinforcing properties of alcohol and decreases drinking motivation and consumption (Viudez-Martínez, García-Gutiérrez, Fraguas-Sánchez, et al., 2018). Further, CBD has shown clinical promise for tobacco, cannabis, and opioid use disorders (Hurd, 2017; Hurd et al., 2015; Prud'homme et al., 2015), and evidence indicates that these effects may be due to the ability of CBD to reduce cue-induced craving and anxiety (Gonzalez-Cuevas et al., 2018; Hurd et al., 2019). The hypotheses are also grounded in the pre-clinical literature suggesting that CBD may modulate the immune system and have anti-inflammatory effects which also helps to reduce harm associated with alcohol and may have a positive effect on those attempting to quit. Other potential mechanisms that might underlie the effects of CBD include a reduction in the severity of acute withdrawal, a reduction in protracted withdrawal, and the neuroprotective effects of CBD. Given the background literature with respect to CBD and AUDs, a logical next step is for human studies to address these questions.

To better understand the effects of hemp-derived CBD with and without a small amount of THC, the investigators propose a Phase II randomized clinical trial (RCT) to examine the safety, tolerability, and clinical effects of Full Spectrum CBD (fsCBD, contains less than 0.3% THC) vs. Broad Spectrum CBD (bsCBD, does not contain THC), vs. a matching placebo in a population of AUD subjects.

This is a double-blind, placebo-controlled, parallel group study designed to assess the efficacy of fsCBD and bsCBD, compared to a placebo control (PC), to reduce drinking in participants with moderate alcohol use disorder according to the DSM-V. If eligible for the study, subjects will be randomized to receive one of the conditions for 8 weeks.

To minimize risk of COVID transmission, the investigators will utilize Zoom for weekly subject check-ins and our Mobile Pharmacology Lab (MPL) for the collection of blood samples and clinical data for the majority of in-person visits. The initial Week 0 / Baseline visit will take place at the University of Colorado Anschutz Medical Campus. There will be MPL follow-up visits at Weeks 1, 4, and 8. Participants will be contacted by Zoom each remaining week during the 8-week period. A follow up Zoom interview will occur in Week 16 approximately 8 weeks after the end of dosing.

Overall, the clinical study is expected to take 1-2 years to complete enrollment and data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between 21-60 years old.
2. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria for current Alcohol Use Disorder (AUD) of at least moderate severity (i.e., 4 or more DSM-V symptoms).
3. Currently seeking treatment for AUD.
4. If male, reports drinking, on average, at least 21 standard alcoholic drinks per week prior to screening; if female, reports drinking, on average, at least 14 standard drinks per week prior to screening.
5. Have at least one heavy drinking day (4 or more drinks per day for women/5 or more drinks per day for men) during the 7-day period prior to screening.
6. Live within 35 miles of the study site.

Exclusion Criteria:

1. Self-reported DSM-V diagnosis of any other substance use disorder.
2. Use nicotine daily.
3. Self-report use of cocaine, amphetamines, opioids, cannabis, or benzodiazepines in the last 30 days.
4. Report having or being treated for a current DSM-V Axis I diagnosis, including major depression, panic disorder, obsessive/compulsive disorder, post-traumatic stress disorder, bipolar affective disorder, schizophrenia, dissociative disorders, eating disorders, or any other psychotic or organic mental disorder.
5. Endorsing an item on the RMTS-S measure of suicide risk.
6. Currently taking any of the following medications:

   1. Those known to have a major interaction with Epidiolex.
   2. Acute treatment with any antiepileptic medications.
   3. Medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, and/or topiramate).
7. Self-reported history of severe alcohol withdrawal (e.g., seizure, delirium tremens).
8. Clinically significant medical problems such as cardiovascular, renal, gastrointestinal, or endocrine problems that would impair participation or limit medication ingestion.
9. Current or past alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, hepatocellular disease, or peptic ulcer.
10. Females of childbearing potential who are pregnant, nursing, or who are not using a reliable form of birth control.
11. Current charges pending for a violent crime (not including DUI-related offenses).
12. Lack of a stable living situation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Drinks per Drinking Day | 0-8 weeks
  The Time Line Follow Back is a calendar-assisted measure that can be used to assess alcohol, tobacco, cannabis, and other substance use. The investigators will use this measure to create the Drinks per Drinking Day variable.
Drinks per Drinking Day | 0-16 weeks
  The Time Line Follow Back is a calendar-assisted measure that can be used to assess alcohol, tobacco, cannabis, and other substance use. The investigators will use this measure to create the Drinks per Drinking Day variable.
Drinks per Drinking Day | 0-4 weeks
  The Time Line Follow Back is a calendar-assisted measure that can be used to assess alcohol, tobacco, cannabis, and other substance use. The investigators will use this measure to create the Drinks per Drinking Day variable.
Drinks per Drinking Day | 4-8 weeks
  The Time Line Follow Back is a calendar-assisted measure that can be used to assess alcohol, tobacco, cannabis, and other substance use. The investigators will use this measure to create the Drinks per Drinking Day variable.
Alcohol Dependence/Craving | 0-16 weeks
  The Alcohol Dependence Scale measures the severity of alcohol dependence. Possible scores range from 0 to 47 with higher scores indicating a worse outcome/more severe symptoms of alcohol dependence. The Penn Alcohol Craving Scale (PACS) measures alcohol craving. Possible scores range from 0 to 30, where higher scores indicate greater craving.
Alcohol Dependence/Craving | 4-8 weeks
  The Alcohol Dependence Scale measures the severity of alcohol dependence. Possible scores range from 0 to 47 with higher scores indicating a worse outcome/more severe symptoms of alcohol dependence. The Penn Alcohol Craving Scale (PACS) measures alcohol craving. Possible scores range from 0 to 30, where higher scores indicate greater craving.
Alcohol Dependence/Craving | 0-8 weeks
  The Alcohol Dependence Scale measures the severity of alcohol dependence. Possible scores range from 0 to 47 with higher scores indicating a worse outcome/more severe symptoms of alcohol dependence. The Penn Alcohol Craving Scale (PACS) measures alcohol craving. Possible scores range from 0 to 30, where higher scores indicate greater craving.
Alcohol Dependence/Craving | 0-4 weeks
  The Alcohol Dependence Scale measures the severity of alcohol dependence. Possible scores range from 0 to 47 with higher scores indicating a worse outcome/more severe symptoms of alcohol dependence. The Penn Alcohol Craving Scale (PACS) measures alcohol craving. Possible scores range from 0 to 30, where higher scores indicate greater craving.

SECONDARY OUTCOMES:
Cue-reactivity | 0-4 weeks
  Cue-elicited urge to drink will be assessed using the cue-reactivity assessment, per protocol (Hutchison, 2006).
Cue-reactivity | 4-8 weeks
  Cue-elicited urge to drink will be assessed using the cue-reactivity assessment, per protocol (Hutchison, 2006).
Cue-reactivity | 0-8 weeks
  Cue-elicited urge to drink will be assessed using the cue-reactivity assessment, per protocol (Hutchison, 2006) .
Anxiety | 0-4 weeks
  The Depression Anxiety and Stress Scale (DASS-21) is a 21-item self-report questionnaire designed to measure three related negative emotional states and yields three subscale scores for depression, anxiety and tension/stress. Possible scores on the anxiety subscale range from 0 to 21, with higher scores indicating more severe symptoms of anxiety.
Anxiety | 4-8 weeks
  The Depression Anxiety and Stress Scale (DASS-21) is a 21-item self-report questionnaire designed to measure three related negative emotional states and yields three subscale scores for depression, anxiety and tension/stress. Possible scores on the anxiety subscale range from 0 to 21, with higher scores indicating more severe symptoms of anxiety.
Anxiety | 0-8 weeks
  The Depression Anxiety and Stress Scale (DASS-21) is a 21-item self-report questionnaire designed to measure three related negative emotional states and yields three subscale scores for depression, anxiety and tension/stress. Possible scores on the anxiety subscale range from 0 to 21, with higher scores indicating more severe symptoms of anxiety.
Anxiety | 0-16 weeks
  The Depression Anxiety and Stress Scale (DASS-21) is a 21-item self-report questionnaire designed to measure three related negative emotional states and yields three subscale scores for depression, anxiety and tension/stress. Possible scores on the anxiety subscale range from 0 to 21, with higher scores indicating more severe symptoms of anxiety.
Subjective Pain Level | 0-4 weeks
  The Adult PROMIS Numerical Rating Scale v1.0 Pain Intensity 1a measures the severity of subjective pain. Possible scores range from 0 to 10, with higher scores indicating more severe symptoms of subjective pain.
Subjective Pain Level | 4-8 weeks
  The Adult PROMIS Numerical Rating Scale v1.0 Pain Intensity 1a measures the severity of subjective pain. Possible scores range from 0 to 10, with higher scores indicating more severe symptoms of subjective pain.
Subjective Pain Level | 0-8 weeks
  The Adult PROMIS Numerical Rating Scale v1.0 Pain Intensity 1a measures the severity of subjective pain. Possible scores range from 0 to 10, with higher scores indicating more severe symptoms of subjective pain.
Subjective Pain Level | 0-16 weeks
  The Adult PROMIS Numerical Rating Scale v1.0 Pain Intensity 1a measures the severity of subjective pain. Possible scores range from 0 to 10, with higher scores indicating more severe symptoms of subjective pain.
Sleep Quality | 0-16 weeks
  The Adult PROMIS Short Form v1.0 Sleep Disturbance 4a measures the severity of sleep disturbances. Possible scores range from 4 to 20, with higher scores indicating more severe symptoms of sleep disturbance.
Sleep Quality | 0-8 weeks
  The Adult PROMIS Short Form v1.0 Sleep Disturbance 4a measures the severity of sleep disturbances. Possible scores range from 4 to 20, with higher scores indicating more severe symptoms of sleep disturbance.
Sleep Quality | 4-8 weeks
  The Adult PROMIS Short Form v1.0 Sleep Disturbance 4a measures the severity of sleep disturbances. Possible scores range from 4 to 20, with higher scores indicating more severe symptoms of sleep disturbance.
Sleep Quality | 0-4 weeks
  The Adult PROMIS Short Form v1.0 Sleep Disturbance 4a measures the severity of sleep disturbances. Possible scores range from 4 to 20, with higher scores indicating more severe symptoms of sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller RL, Hooper JF, Ellingson JM, Olsavsky AK, Rzasa-Lynn R, Bryan AD, Bidwell LC, Hutchison KE. A preliminary randomized trial of the safety, tolerability, and clinical effects of hemp-derived cannabidiol in alcohol use disorder. Front Psychiatry. 2025 Apr 28;16:1516351. doi: 10.3389/fpsyt.2025.1516351. eCollection 2025. PMID 40357520